CLINICAL TRIAL: NCT05271318
Title: A Two-part, Phase I/Ib, Open-Label, Dose-escalation Trial of Tumor Necrosis Factor Alpha and Interleukin-2 Coding Oncolytic Adenovirus (TILT-123) in Combination With Pembrolizumab (Phase I Part) and Pembrolizumab and Pegylated Liposomal Doxorubicin (Phase Ib Part) in Patients With Platinum Resistant or Refractory Ovarian Cancer
Brief Title: Oncolytic Adenovirus Coding for TNFa and IL2 (TILT-123) With Pembrolizumab or Pembrolizumab (Phase 1a) and Pegylated Liposomal Doxorubicin (Phase 1b) as Treatment for Ovarian Cancer.
Acronym: PROTA
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: TILT Biotherapeutics Ltd. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TILT-T563; OC220391 (Other Grant/Funding Number: US Department of Defense); 2021-005083-22 (EudraCT Number); MK-3475-C70 (Other: Merck Sharp & Dohme LLC); KEYNOTE-C70 (Other: Merck Sharp & Dohme LLC)
Record Dates: First submitted 2022-02-04; First posted 2022-03-09 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Platinum-refractory Ovarian Carcinoma; Platinum-resistant Ovarian Cancer; Platinum-Resistant Fallopian Tube Carcinoma; Platinum-Resistant Primary Peritoneal Carcinoma; Platinum-Refractory Fallopian Tube Carcinoma; Platinum-Refractory Primary Peritoneal Carcinoma; Platinum-Sensitive Ovarian Cancer in Which the Participant Has Allergy or Severe Intolerance to Carboplatin and/or Cisplatin; Platinum-Sensitive Fallopian Tube Carcinoma in Which the Participant Has Allergy or Severe Intolerance to Carboplatin and/or Cisplatin; Platinum-Sensitive Primary Peritoneal Carcinoma in Which the Participant Has Allergy or Severe Intolerance to Carboplatin and/or Cisplatin
Keywords: Oncolytic virus; Virotherapy; Immune checkpoint inhibitor; Adenovirus; TILT-123; Pembrolizumab; anti-Programmed Cell Death 1 (anti-PD1); Keytruda
MeSH Terms: conditions — Adenoviridae Infections | interventions — pembrolizumab; liposomal doxorubicin; 1-dodecylpyridoxal

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1 part - TILT-123 and pembrolizumab (Experimental): Patients will receive multiple administrations of TILT-123 and pembrolizumab.
  Escalation to the next dose of TILT-123 level will occur when the safety data has been evaluated for all patients in the preceding dose level.
  Interventions: Biological: TILT-123; Biological: pembrolizumab
- Phase 1b part - TILT-123 and pembrolizumab and pegylated liposomal doxorubicin (Experimental): Patients will receive multiple administrations of TILT-123 and pembrolizumab and pegylated liposomal doxorubicin.
  TILT-123 will be administered at the maximum tolerated dose or maximum feasible dose.
  Interventions: Biological: TILT-123; Biological: pembrolizumab; Drug: pegylated liposomal doxorubicin

INTERVENTIONS:
Biological: TILT-123 — Tumor necrosis factor alpha (TNFalpha) and Interleukin-2 (IL-2) coding oncolytic adenovirus TILT-123
  Other Names: Ad5/3-E2F-d24-hTNFa-IRES-hIL2 (TILT-123)
Biological: pembrolizumab — pembrolizumab, a monoclonal antibody binding PD-1
  Other Names: KEYTRUDA®; MK-3475
Drug: pegylated liposomal doxorubicin — Pegylated Liposomal Doxorubicin is a chemotherapy and a pegylated liposomal form of the anthracycline topoisomerase inhibitor, doxorubicin.
  Other Names: PLD
  Arms: Phase 1b part - TILT-123 and pembrolizumab and pegylated liposomal doxorubicin

SUMMARY:
This is an open-label, phase 1/1b, dose-escalation, multicenter and multinational trial evaluating the safety of oncolytic adenovirus TILT-123 in combination with Pembrolizumab, or Pembrolizumab and Pegylated Liposomal Doxorubicin in patients with platinum resistant or refractory ovarian cancer.

DETAILED DESCRIPTION:
This is an open-label, phase 1/1b, dose-escalation, multicenter and multinational trial evaluating the safety of oncolytic adenovirus TILT-123 in combination with Pembrolizumab, or Pembrolizumab and Pegylated Liposomal Doxorubicin in patients with platinum resistant or refractory ovarian cancer. TILT-123 is an oncolytic adenovirus coding for tumor necrosis factor alpha (TNFa) and interleukin 2 (IL-2). Pembrolizumab is a monoclonal antibody binding program cell death 1 (PD-1). Pegylated Liposomal Doxorubicin is a chemotherapy and a pegylated liposomal form of the anthracycline topoisomerase inhibitor, doxorubicin.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent(s) by the participant or legal representative before any trial-related activities.
* Female over 18 years of age on day of signing informed consent(s).
* Diagnosis:

  1. Phase I part: Histologically confirmed ovarian cancer (including fallopian tube and primary peritoneal cancer) resistant to platinum (defined as progression of cancer within 183 days of the most recent dose of cisplatin or carboplatin) or refractory to platinum (defined as progression of cancer within 30 days of the most recent dose of cisplatin or carboplatin) ovarian cancer, which cannot be treated with curative intent with available therapies.
  2. Phase Ib part: Platinum refractory/resistant ovarian cancer treated with up to one line of prior chemotherapy in refractory/resistant setting. Note: A regimen that contains only one or more biological agents and/or targeted therapies but no cytotoxic drug does not count as a line of chemotherapy Note: For both phase I and phase Ib, PARP inhibitors should be considered as indicated in clinical practice, prior to trial enrollment. Patients who have platinum-sensitive disease (no recurrence or progression within 183 days of the last dose of platinum-containing chemotherapy) but who have an allergy or severe intolerance to carboplatin and/or cisplatin may be included.
* At least one tumor (>14 mm in diameter) or carcinomatosis must be available for local virus injection (intratumoral and/or intraperitoneal).
* The disease burden must be evaluable, but does not need to fulfil RECIST 1.1.
* Have adequate organ function as defined in the following values below. Specimens must be collected within 10 days prior to the start of study treatment.

  a. Hematological laboratory values i. Absolute neutrophil count (ANC): ≥1500/µL ii. Platelets: ≥ 100 000/µL iii. Hemoglobin: ≥9.0 g/dL or ≥5.6 mmol/L. Criteria must be met without packed red blood cell (pRBC) transfusion within the prior 2 weeks. Participants can be on stable dose of erythropoietin (≥ approximately 3 months. iv. Leukocytes (WBC) > 3.0x10^9/L b. Renal laboratory values i. Glomerular Filtration Rate (GFR): >45 ml/min (CKD-EPI formula). c. Hepatic laboratory values i. Total bilirubin: ≤1.5 × Upper Limit of Normal (ULN) OR direct bilirubin ≤ULN for participants with total bilirubin levels >1.5 × ULN (excluding patients with Gilber's Disease) ii. Aspartate Aminotransferase (AST) (SGOT) and Alanine Aminotransferase (ALT) (SGPT): ≤2.5 × ULN (≤5 × ULN for participants with liver metastases)
* Patients must be willing to use adequate forms of contraception from screening, during the trial, and for a minimum of 120 days after end of treatment, in accordance with the following:

  i. Women of childbearing potential: Barrier contraceptive method (i.e. condom) must be used in addition to one of the following methods: Intrauterine devices or hormonal contraception (oral contraceptive pills, implants, transdermal patches, vaginal rings or long-acting injections). ii. Women not of childbearing potential: Barrier contraceptive method (i.e. condom) must be used.
* Eastern Cooperative Oncology Group (ECOG)/World Health Organization (WHO) performance score of 0-1 at screening.
* Life expectancy longer than 3 months.
* Capable of understanding and complying with parameters as outlined in the protocol.

Exclusion Criteria:

* Has an active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) and inhaled and topical treatments are not considered a form of systemic treatment and are allowed.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior the first dose of study drug.
* Prior therapy:

  1. Both phase I and phase Ib parts: Treated with any anti-cancer therapy within 30 days prior to the first virus injection. Anti-cancer therapy is defined as anti cancer agents (e.g. surgery, chemotherapy, immune-checkpoint inhibitors, kinase inhibitors, PARP inhibitors, biological therapies, hormonal therapies, radiation, etc.). Continuation of hormonal therapy or use of bone modifying agents (e.g. bisphosphonate or denosumab) is allowed if started at least 3 months before.
  2. Phase Ib part: Prior oncolytic viruses, immune checkpoint inhibitors or anthracyclines (eg. doxorubicin, liposomal doxorubicin, epirubicin or any other anthracycline formulations).
* Participants must have recovered from all Adverse Events (AE)s due to previous therapies to ≤Grade 1or baseline. Participants with ≤Grade 2 neuropathy may be eligible. Participants with endocrine-related AEs Grade ≤2 requiring treatment or hormone replacement may be eligible. If the participant had major surgery, the participant must have recovered adequately from the procedure and/or any complications from the surgery prior to starting study intervention.
* Treated with a prior radiotherapy, including for palliative purposes, within 2 weeks of start of study treatment (before or after). Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-Central Nervous System (CNS) disease. Palliative radiation is allowed from day 15 during the trial treatment period, if deemed necessary by the investigator.
* Treated with a prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., Cytotoxic T lymphocyte-associated Antigen (CTLA)-4, Tumor necrosis factor receptor superfamily, member 4 (OX40), CD137), and was discontinued from that treatment due to a Grade 3 or higher immune-related Adverse Events (irAE).
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 30 days prior to the first virus injection. An investigational agent is any drug or therapy that is currently not approved for use in humans. Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.
* Uncontrolled cardiac or vascular diseases.
* History of myocardial infarction or cerebral stroke within the previous 12 months before screening or is not sufficiently recovered from an older infarction or cerebral stroke.
* History of severe hepatic dysfunction.
* History of hepatitis B (defined as HBsAg reactive), Hepatitis C (defined as hepatitis C virus (HCV) RNA [qualitative] is detected) and/or HIV. No testing for Hepatitis B, Hepatitis C and HIV is required unless mandated by a local health authority.
* History of coagulation disorder.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating investigator.
* Female patients who are pregnant, breastfeeding or intend to become pregnant. Women of childbearing potential who has a positive urine pregnancy test (within 72 hours) prior to treatment. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Has a known additional malignancy that is progressing or has required active treatment within the past 5 years. Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g., breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.
* Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e., without evidence of progression for at least 3 months by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment.
* Has an active infection requiring systemic therapy.
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
* Has a known psychiatric or substance abuse disorder that would interfere with the participant's ability to cooperate with the requirements of the study.
* Allergy to ingredients present in the investigational medicinal products (ingredients are listed in the protocol) ie. severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
* Known contraindications to pembrolizumab.
* Has had an allogenic tissue/solid organ transplant.
* Has received a live or live-attenuated vaccine within 30 days prior to the first dose of study intervention. Administration of killed vaccines are allowed.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2022-05-17 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with any (serious and non-serious) Adverse Events | Day 92
Number of Participants with vital sign abnormalities | Day 92
Number of Participants with abnormal laboratory values | Day 92
Number of Participants with Adverse Events assessed by electrocardiograms (ECGs) | Day 92

CONTACTS AND LOCATIONS:
Locations (3):
- United States (2):
  - Mayo Clinic, Rochester, Minnesota
  - Northwell Heatlh/Lenox Hill Hospital, New York, New York
- Docrates Cancer Center, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Havunen R, Kalliokoski R, Siurala M, Sorsa S, Santos JM, Cervera-Carrascon V, Anttila M, Hemminki A. Cytokine-Coding Oncolytic Adenovirus TILT-123 Is Safe, Selective, and Effective as a Single Agent and in Combination with Immune Checkpoint Inhibitor Anti-PD-1. Cells. 2021 Jan 27;10(2):246. doi: 10.3390/cells10020246. PMID 33513935
- [Background] Cervera-Carrascon V, Siurala M, Santos JM, Havunen R, Tahtinen S, Karell P, Sorsa S, Kanerva A, Hemminki A. TNFa and IL-2 armed adenoviruses enable complete responses by anti-PD-1 checkpoint blockade. Oncoimmunology. 2018 Apr 9;7(5):e1412902. doi: 10.1080/2162402X.2017.1412902. eCollection 2018. PMID 29721366
- [Derived] Clubb JHA, Pakola SA, Joenvaara S, Kudling TV, Tohmola T, Arias V, Jirovec E, van der Heijden M, Quixabeira DCA, Pasanen A, Haybout L, Ojala N, Basnet S, Eleuteri A, Ferrero JD, Hirvenoja S, Svane IM, Maenpaa J, Jalkanen K, Block MS, Alanko T, Monberg T, Zahraoui S, Gronberg-Vaha-Koskela S, Salmelin N, Kistler C, Havunen R, Sorsa S, Manuel Dos Santos J, Cervera-Carrascon V, Kanerva A, Hemminki O, Renkonen R, Hemminki A. Dyslipidemia-associated natural IgM improves oncolytic virus TILT-123 efficacy through antibody-dependent enhancement in solid tumors. Mol Ther. 2026 Jan 20:S1525-0016(26)00020-1. doi: 10.1016/j.ymthe.2026.01.019. Online ahead of print. PMID 41566775
- [Derived] Jirovec E, Quixabeira DCA, Clubb JHA, Pakola SA, Kudling T, Arias V, Haybout L, Jalkanen K, Alanko T, Monberg T, Khammari A, Dreno B, Svane IM, Block MS, Adamo DA, Maenpaa J, Kistler C, Sorsa S, Hemminki O, Kanerva A, Santos JM, Cervera-Carrascon V, Hemminki A. Single intravenous administration of oncolytic adenovirus TILT-123 results in systemic tumor transduction and immune response in patients with advanced solid tumors. J Exp Clin Cancer Res. 2024 Nov 6;43(1):297. doi: 10.1186/s13046-024-03219-0. PMID 39506856